CLINICAL TRIAL: NCT02064088
Title: Volume or Concentration for the Transverse Abdominal Plane Block in Children Aged 1-5 Years: Analgesic Effects and Safety
Brief Title: Transversus Abdominis Plane Block in Pediatrics: Volume or Concentration ?
Acronym: TAP Bloc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UF9206
Record Dates: First submitted 2014-02-04; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Inguinal or Ovarian Hernia; Hydrocele; Cord Kyst; Local Analgesia Block; One to Five Years
Keywords: Regional anesthesia; TAP block; Pediatric anesthesia; analgesic effects; pharmacokinetics
MeSH Terms: conditions — Testicular Hydrocele

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Small volume (Experimental): Local analgesia by one injection of 0,2 ml/kg of 0,2% lévobupivacaine
  Interventions: Drug: Injection of 0,2 ml/kg of 0,2% levobupivacaine for small volume group
- High volume (Experimental): Local analgesia by one injection of 0,4 ml/kg of 0,1% lévobupivacaine
  Interventions: Drug: Injection of 0,4 ml/kg of 0,1% lévobupivacaine for high volume group

INTERVENTIONS:
Drug: Injection of 0,2 ml/kg of 0,2% levobupivacaine for small volume group — Ultrasound guided administration of 0,2 ml/kg of 0,2% lévobupivacaine in the plane between the internal oblique and transversus abdominis muscles
  Arms: Small volume
Drug: Injection of 0,4 ml/kg of 0,1% lévobupivacaine for high volume group — Ultrasound guided administration of 0,4 ml/kg of 0,1% lévobupivacaine in the plane between the internal oblique and transversus abdominis muscles
  Arms: High volume

SUMMARY:
The transversus abdominis plane (TAP) block provide a local anesthesia drug diffusion between the transverse abdominis muscle and the internal oblique muscle. TAP block reaches the anterior rami of spinal nerves from T7 to L1 involved in the innervation of homolateral abdominal wall. The transversus abdominis plane block has shown promise for perioperative analgesia, but data on the optimal dose regimen are limited.Following previous research of optimal dose of local anesthesic solution, the investigators aim to evaluate if a "volume effect" would lead to a better diffusion of the local anesthesic solution to the overall nervous roots. The local anesthesia drug choosen is levobupivacaine with a unique posology of 0,4 mg/kg (either 0,2 ml/kg of 0,2% levobupivacaine for "small volume" group or 0,4 ml/kg of 0,1% levobupivacaine for "high volume" group).With the same dose of levobupivacaine, this study aims to assess the impact of volume effect on analgesia efficiency as well as the security as after ultrasound TAP block on one to five years' old children who undergo a peritoneal-vaginal duct surgery.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation in ambulatory surgery and anesthesia unit for surgery of inguinal hernia or ovarian hernia or hydrocele or cord kyst
* Overall status: ASA I-II
* Aged from 1 to 5 years
* Informed consent

Exclusion Criteria:

* Coagulation trouble
* Infection on ponction zone
* Local anesthesia drug or nonsteroidal anti inflammatory intolerance
* Cardiac/Renal/hepacticdysfunction
* Hemorrage, digestive perforation history

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
number of patients for whom a rescue analgesia was necessary in post anesthesia care unit and ambulatory surgery unit | from arrival in post anesthesia care unit until discharge (An expected average of 4 hours after end of surgery)

SECONDARY OUTCOMES:
Intraoperative opioid consumption : total Rémifentanil (µg/kg) | for time of surgery (1 to 4 hours)
Post operative pain (FLACC scale) at hospital | from recovery room until discharge (An expected average of 4 hours after end of surgery)
  Post operative pain is evaluated every 15 minutes in the recovery room and then every two hours in the ambulatory surgical unit until discharge at home.
Plasmatique peak of levobupivacaine (Cmax in µg/ml) | 5 min until 75 min after injection of local anaesthetic
Time necessary to reach plasmatique peak of levobupivacaine (tmax in min) | 5 min until 75 min after injection of local anaesthetic
Complications related to local analgesia procedure | until 24 hours in post operative
  cardiovascular adverse event, adverse vascular ponction (positive aspiration test for blood), adverse peritoneal ponction, hematoma
First request of rescue antalgic (Nubain or Tramadol) | until 24 hours in post operative
Consommation of rescue antalgic | until 24 hours in post operative
Pain evaluation at home by parents (score PPMP) | call between 24 and 48 hours in post operative

CONTACTS AND LOCATIONS:
Overall Officials: Chrystelle CS SOLA, MD, Principal Investigator — CHU Montpellier - Lapeyronie Hospital
Locations (1):
- CHU Montpellier, Montpellier, France

REFERENCES:
- [Derived] Sola C, Menace C, Bringuier S, Saour AC, Raux O, Mathieu O, Capdevila X, Dadure C. Transversus Abdominal Plane Block in Children: Efficacy and Safety: A Randomized Clinical Study and Pharmacokinetic Profile. Anesth Analg. 2019 Jun;128(6):1234-1241. doi: 10.1213/ANE.0000000000003736. PMID 31094793